CLINICAL TRIAL: NCT06486051
Title: A Phase 2 Trial to Evaluate the Efficacy and Safety of WZTL-002 in Patients With Relapsed or Refractory Large B-cell Lymphoma (ENABLE-2)
Brief Title: A Study of WZTL-002 CAR T-cells for Adults With Relapsed Large B-cell Lymphoma
Acronym: ENABLE-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Malaghan Institute of Medical Research (Other)
Collaborators: BioOra Limited (Unknown); Wellington Zhaotai Therapies Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WZTL002-2; U1111-1305-7917 (Other: World Health Organization)
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Large B-cell Lymphoma; Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Primary Mediastinal Large B-cell Lymphoma (PMBCL); Transformed Non-Hodgkin Lymphoma
Keywords: Chimeric Antigen Receptor Therapy; CD19 Antigen; Toll-Like Receptor 2; CD28 Antigen; Relapsed non-Hodgkin Lymphoma; Refractory non-Hodgkin Lymphoma; Adoptive Cellular Immunotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WZTL002 CAR T-cells (Experimental): Target dose of 0.85×10^6 CAR+ cells per kg body weight (target range 0.5 to 1.0×10^6 CAR+ cells/kg; dose cap 1×10^8 cells)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: WZTL-002 CAR T-cells

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m^2/day IV for three consecutive days
Drug: Cyclophosphamide — 500 mg/m^2/day IV for three consecutive days
Biological: WZTL-002 CAR T-cells — WZTL-002 comprises autologous T-cells transduced to express the third-generation 1928T2z chimeric antigen receptor, which recognises the CD19 antigen present on malignant and normal B-cells. The chimeric antigen receptor (CAR) incorporates an extracellular scFv specific for CD19, the intracellular signalling domains of CD28 and CD3ζ, and an intracellular co-stimulatory domain derived from TLR2 interposed between CD28 and CD3ζ.
  On Day 0, the WZTL-002 CAR T-cell product is administered intravenously two days after completing lymphodepleting chemotherapy.
  Other Names: 1928T2z CAR T-cells

SUMMARY:
The goal of this clinical trial is to learn if a new type of chimeric antigen receptor (CAR) T-cell therapy called WZTL-002 is effective and safe for the treatment large B-cell lymphomas (LBCL) that have not responded to or have come back after standard chemotherapy. The main questions this trial aims to answer are:

* What is the likelihood of complete response of the lymphoma after WZTL-002 treatment?
* What is the risk of altered brain function (neurotoxicity) after WZTL-002?

All eligible participants will receive WZTL-002; the researchers will compare the complete response rate and neurotoxicity rate with historical groups of patients who were treated with similar therapies.

Participants will:

* Have a procedure to gather white blood cells
* Receive chemotherapy to prepare for the CAR T-cells
* Receive WZTL-002 CAR T-cells through a vein
* Be monitored closely for the first 14 days for certain side effects
* Have scans 28 days and 3, 6, 12 and 24 months after WZTL-002 CAR T-cells to check if the treatment has worked

DETAILED DESCRIPTION:
WZTL-002 is a third-generation CAR T-cell product comprising autologous T-cells transduced to express a CAR directed against CD19 and incorporating a Toll-like receptor 2 (TLR2) co-stimulatory domain interposed between CD28 and CD3ζ signalling domains. The trial will screen up to 80 patients in order to enrol and treat approximately 60 participants with WZTL-002. This is a single arm open-label phase 2 trial designed to evaluate the efficacy, safety, cellular kinetics and pharmacodynamic properties of WZTL-002 for the second- or third-line treatment of r/r LBCL.

Eligible participants will undergo leukapheresis to harvest peripheral blood mononuclear cells, the starting material for the manufacture of the autologous third generation anti-CD19 CAR T-cell product, WZTL-002. After WZTL-002 manufacture and confirmation that product release criteria are met, participants will receive lymphodepleting chemotherapy comprising fludarabine and cyclophosphamide on days -5 to day -3, inclusive. WZTL-002 will be administered intravenously on day 0 as a single dose.

After WZTL-002 administration, participants will be monitored closely for 14 days including targeted assessments for the specific CAR T-cell related toxicities Cytokine Release Syndrome (CRS) and Immune Effector Cell Neurotoxicity Syndrome (ICANS). CRS, ICANS and grade 3 or higher neutropenia, thrombocytopenia or anemia persisting beyond day 30 will be recorded as adverse events of special interest. PET/CT scans to assess treatment response will take place at screening, pre-lymphodepletion and at 28 days, 3 months and 6 months after WZTL-002 infusion, and CT scans to assess duration of response at 12 and 24 months after WZTL-002 infusion. Samples will be taken to determine WZTL-002 cellular kinetics and the depth and duration of B-cell aplasia (pharmacodynamic analysis).

Follow-up beyond month 24 will take place within the Center for International Blood and Marrow Transplant Research (CIBMT) Cellular Therapies Registry or the Australasian Bone Marrow Transplant Recipient Registry (ABMTRR), and in a subsequent long-term follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years (inclusive) at the time of informed consent
2. Signed written informed consent for this trial
3. Biopsy-proven relapsed or treatment-refractory B-cell non-Hodgkin lymphoma of the following subtypes, as per the 2022 WHO classification of haematolymphoid tumours

   * Large B-cell lymphomas of the following histological subtypes:

     * Diffuse LBCL, not otherwise specified
     * Diffuse large B-cell lymphoma/high grade B-cell lymphoma with MYC and BCL2 rearrangements
     * Large B-cell lymphoma with IRF4 rearrangement
     * High grade B-cell lymphoma with 11q aberrations
     * High grade B-cell lymphoma, not otherwise specified
     * Primary mediastinal large B-cell lymphoma
     * Follicular large B-cell lymphoma
     * EBV-positive diffuse large B-cell lymphoma, not otherwise specified
     * Diffuse large B-cell lymphoma associated with chronic inflammation
     * Primary cutaneous DLBCL, leg type
   * Large B-cell lymphoma of one of the above subtypes that has transformed from follicular or marginal zone lymphoma
4. Received adequate first-line lymphoma therapy for the qualifying histology (as defined in inclusion criterion 3 above), comprising at least 2 cycles of a standard combination regimen incorporating an anthracycline and an anti-CD20 monoclonal antibody
5. Relapsed or refractory disease meeting one of the following criteria:

   * Relapsed or refractory within 12 months of first-line chemoimmunotherapy, defined as:

     * Progressive disease following ≥ 2 cycles of chemoimmunotherapy, or
     * Stable disease following ≥ 4 cycles of chemoimmunotherapy, or
     * Partial response following ≥ 6 cycles of chemoimmunotherapy, or
     * Complete response followed by biopsy-proven relapse within 12 months of completing first-line chemoimmunotherapy.
   * Relapsed or refractory following second-line chemoimmunotherapy, defined as:

     * Lack of complete response to, or relapse following, autologous stem cell transplantation as part of second-line therapy for the qualifying histology, or
     * Inability to proceed to autologous stem cell transplantation due to lack of response to 2 cycles of second-line chemoimmunotherapy incorporating both a platinum agent and an anti-CD20 monoclonal antibody
6. Positron emission tomography (PET) positive disease according to the Lugano 2014 criteria
7. Available tumour tissue (comprising a tissue block or at least 6 unstained slides) for central histological review
8. Lymphoma-related life expectancy at least 12 weeks, and life expectancy related to conditions other than lymphoma at least 12 months
9. ECOG performance status of 0 or 1
10. Adequate haematologic function, defined by:

    * Neutrophils ≥ 1.0 × 10^9/L, and Platelets ≥ 75 × 10^9/L, and
    * Lymphocytes ≥ 0.3 × 10^9/L
11. Adequate renal function, defined by estimated creatinine clearance (eCrCl) or glomerular filtration rate (eGFR) >/= 45mL/min using the Cockroft Gault estimation, CKD-EPI equation or as assessed by direct measurement.
12. Adequate hepatic function, defined by serum bilirubin < 2.5 × upper limit of normal (ULN) (unless attributable to Gilbert's syndrome) and alanine transaminase and aspartate aminotransferase < 3 × ULN.
13. Adequate lung function, defined as ≤ Grade 1 dyspnoea according to NCI CTCAE v5.0, and oxygen saturation (sO2) ≥ 92% on room air.
14. Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) ≥ 40% as assessed by echocardiogram or multigated acquisition (MUGA), performed within 28 days of commencing screening.
15. For female participants:

    * Agree to use a condom if undertaking sexual activity with any partner during lymphodepleting chemotherapy, and
    * If of reproductive potential agree to use a highly effective method of contraception from the time of enrolment until at least 12 months after administration of WZTL-002, or
    * Are not of reproductive potential defined as either,

      * being amenorrhoeic for at least 12 consecutive months with FSH 30 ≥ IU/L, or
      * previously undergone a sterilisation procedure
16. For male participants:

    * Agree to use a condom if undertaking sexual activity with any partner during lymphodepleting chemotherapy, and
    * If undertaking sexual activity with a female partner of reproductive potential agree to use a highly effective method of contraception from the time of enrolment until at least 12 months after administration of WZTL-002, and
    * Agree not to donate sperm for conception, or to provide gametes for in vitro fertilisation for at least 12 months after administration of WZTL-002
17. Participant agrees not to donate blood components at any time after receiving WZTL-002

Exclusion Criteria:

1. Active central nervous system (CNS) involvement by lymphoma. In patients with a history of CNS disease or a clinical suspicion of current CNS disease, lumbar puncture and MRI brain must be performed within 30 days of enrolment to exclude current CNS involvement.
2. Active CNS pathology including: epilepsy, seizure within the preceding year, aphasia, paresis, stroke, dementia, psychosis within the preceding year, severe brain injury, Parkinson disease, or cerebellar disease
3. B-cell non-Hodgkin lymphoma of the following subtypes, as per the 2022 WHO classification of haematolymphoid tumours:

   * Richter transformation of chronic lymphocytic leukaemia
   * T-cell/histiocyte rich LBCL
   * Primary LBCL of immune-privileged sites
   * Fluid overload associated LBCL
   * Fibrin-associated LBCL
   * Plasmablastic lymphoma
   * Mediastinal grey zone lymphoma
   * Intravascular LBCL
   * ALK-positive large B-cell lymphoma
   * Lymphomatoid granulomatosis
   * Burkitt lymphoma
   * Primary effusion lymphoma
   * KSHV/HHV8-positive diffuse large B-cell lymphoma
4. Patient has received 3 or more prior lines of therapy for LBCL, where 1 line of therapy is defined as 1 or more cycles of a combination chemoimmunotherapy with or without pre-planned consolidation therapy (radiotherapy, autologous stem cell transplant or immunotherapy)
5. Requirement for urgent lymphoma therapy due to tumour-related symptoms, or due to imminent risk of blood vessel, airway, urinary tract, gastrointestinal tract, nerve or spinal cord compression
6. Active autoimmune disease requiring current systemic immunosuppression
7. Active sarcoidosis
8. Prior solid organ transplantation or prior allogeneic stem cell transplantation (allo-SCT)
9. Peripheral blood CD3+ T cells < 150/μL (0.15 x10^9/L) as assessed by lymphocyte subset analysis
10. History of active malignancy other than B-cell malignancy within 2 years prior to enrolment, with the exception of: adequately treated in situ carcinoma of the cervix; adequately treated basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) of the skin; other localised malignancy surgically resected (or radically treated with another treatment modality) with curative intent
11. Prior treatment with:

    * gene therapy (including CAR T-cell therapy) or CD19-targeted immunotherapy, or
    * purine analogue (including bendamustine) or alemtuzumab within 6 months of enrolment, or
    * bispecific T-cell engager, radiotherapy or an investigational medicine within 4 weeks of enrolment, or
    * cytotoxic chemotherapy, systemic corticosteroids (at doses of ≥ 10 mg prednisone daily or equivalent), monoclonal antibody or antibody-drug conjugate (other than alemtuzumab) within 2 weeks of enrolment.
12. Pregnant or lactating female
13. Known sensitivity to immunoglobulin or to components of the IP
14. Current or prior HIV infection
15. Vaccination with a live virus within the 4 weeks of enrolment
16. Inadequately-controlled systemic infection
17. Serologic status reflecting active viral hepatitis B or active hepatitis C infection as follows:

    * Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Patients with presence of HBcAb, but absence of HBsAg, are eligible if hepatitis B virus (HBV) DNA is undetectable (or is < 20 IU/mL), and if they are willing to receive appropriate antiviral prophylaxis.
    * Presence of active Hepatitis C infection as determined by Hepatitis C virus (HCV) RNA detected by PCR or nucleic acid testing (NAT). Patients with presence of HCV antibody, are eligible if HCV RNA is undetectable.
18. Current New York Heart Association (NYHA) class 2 or higher cardiac symptoms, or myocardial infarction, unstable angina or other clinically significant cardiac disease within the past 6 months
19. Significant concomitant illnesses which would in the Investigators opinion make the patient an unsuitable candidate for the trial
20. Patients who have diminished capacity or any circumstance that would prohibit them from understanding and providing informed consent in accordance with ICH-GCP
21. Patient does not provide consent to enrol to an International Cellular Therapy Registry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate per Investigator assessment | 3 months after WZTL-002 administration
  Investigator-assessed CR rate according to Lugano Response Criteria
Immune effector cell-associated neurotoxicity syndrome (ICANS) rate | 3 months after WZTL-002 administration
  Proportion of participants with ICANS (any grade) as assessed by American Society for Transplantation and Cellular Therapy (ASTCT) criteria

SECONDARY OUTCOMES:
Complete response (CR) rate per central assessment | 3 months after WZTL-002 administration
  Complete response (CR) rate per central assessment according to Lugano Response criteria
Objective response rate (ORR) per investigator and per central assessment | At 3 and at 6 months after WZTL-002 administration
  Objective response rate comprising CR rate plus partial response (PR) rate, according to Lugano Response Criteria
Progression free survival (PFS), Event-free survival (EFS), Overall survival (OS) and Duration of Response (DOR) | At Months 3, 6, 9, 12, 18, and 24 after WZTL-002 administration
  To estimate the progression-free, event-free, overall survival and duration of response after treatment with WZTL-002
Cytokine release syndrome (CRS) rate and grade | 3 months after WZTL-002 administration
  CRS rate and grade, as assessed by ASTCT consensus criteria
Number and severity of adverse effects | From screening until 24 months after WZTL-002 administration
  Adverse events will be graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria (except for CRS and ICANS; see separate endpoints)
Hospitalisation (inpatient) days | 3 months after WZTL-002 administration
  Number of intensive care unit (ICU) inpatient days and non-ICU inpatient days and reason for hospitalisation
Health-related quality of life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Upto 24 months after WZTL-002 administration
  EORTC QLQ-C30 is a 30-item participant self-reported questionnaire composed of multi-item and single scales. Participants rate items and a score from 0 to 100 for the global health status scale and for each functional scale is calculated. A higher score indicates a better level of quality of life or function, and positive changes from baseline indicate improvement
European Quality of Life 5-Dimensions 5-Levels Health Questionnaire (EQ-5D-5L) | Upto 24 months after WZTL-002 administration
  The EQ-5D-5L measures health outcomes using a visual analogue score (VAS) to record a participant's self-rated health on a scale from 0 to 100, where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine.' A higher score indicates a better health outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Philip George, MBChB, Principal Investigator — Te Whatu Ora Health New Zealand, Capital Coast & Hutt Valley; Robert Weinkove, PhD, Study Chair — Malaghan Institute of Medical Research
Locations (3):
- New Zealand (3):
  - Christchurch Hospital, Christchurch, Christchurch Central
  - Wellington Hospital, Newtown, Wellington Region
  - Auckland City Hospital, Auckland

IPD SHARING:
Plan to Share IPD: No